CLINICAL TRIAL: NCT04410705
Title: Investigation the Effect of the Extracorporeal Shock Wave Therapy on Muscle Strength, Flexibility and Architectural Features in Lower Extremity Tendinopathies
Brief Title: Effect of Eswt on Muscle Architecture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aydan Niziplioğlu, MSc. physiotherapist, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01
Record Dates: First submitted 2020-05-11; First posted 2020-06-01 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Tendinopathy
Keywords: Extracorporeal shockwave theraphy; Ultrasonography; muscle strength
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Intervention Model Description: ESWT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tendinopathy patients (Experimental): Patients with tendinopathy will be administered ESWT
  Interventions: Other: Extracorporeal shockwave theraphy for hamstring tendinopathy; Other: Extracorporeal shockwave theraphy for quadriceps tendinopathy; Other: Extracorporeal shockwave theraphy for achilles tendinopathy

INTERVENTIONS:
Other: Extracorporeal shockwave theraphy for hamstring tendinopathy — For hamstring tendinopathy; a total of 2000 impulses will be done. We will apply twice a week and 5 times in total.
Other: Extracorporeal shockwave theraphy for quadriceps tendinopathy — Energy flux density will be 0.58mJ/mm2 (2 bar) with 2000 impulses. We will perform twice a week, 5 times in total.
Other: Extracorporeal shockwave theraphy for achilles tendinopathy — Each session consisted of 2400 impulses will be administered with an energy flux density ranged from 0.17 to 0.25 mJ/mm2 (1.7-2.5 bar). We will perform once a week, 3 times in total.

SUMMARY:
The aim of the research is to investigate the effect of Ekstracorpereal shock wave treatment (ESWT) on muscle strength, flexibility and architecture of the lower extremity tendinopathies when applied using the frequencies specified in the literature with min and max frequency frequencies.

Our hypothesis as researchers is ESWT treatment has an effect on muscle strength, flexibility and muscle architecture.

DETAILED DESCRIPTION:
The study will conduct in the Physical Therapy and Radiology Department in a private hospital. The Clinical Research Ethics Committee of Gaziantep the univsersity approved ethical compliance of the study with the decision number GO 2018-01. The participants will inform about the study and their write consent will obtain.

Demographic information including the name, age, height, body weight and occupation of the participants will obtain before the evaluation. All the measurements will perform before, soon after the 1st session and after the last session.

Outcome measures will be muscle strength, muscle flexibility, muscle architectures parameters.

ELIGIBILITY:
Inclusion Criteria: Lower extremity tendinopathy

Exclusion Criteria:

* Patients who failed to show up to any treatment and measurement sessions,
* Patients who cannot tolerate treatment
* having systemic inflammatory disease,
* lower or upper motor lesion

Ages: 21 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-07-05 (Actual); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
muscle pannation angle | Measurements will perform prior to ESWT,immidiately after the first ESWT and last ESWT treatment. Change of pannation angle in 3 weeks
  'Logiq s7 Expert' US device including b-flow, semi-quantification and elastography, flow quantification, contrast imaging, b-steer and volume imaging device and with 11 L-D linear volume convex and linear probe will use for the measurements. During the evaluation, the muscles will place in the most relaxed position and no contraction will request. Pennation angle will measure as the angle between muscle fibre and the deep fascia of the muscle
muscle fiber length | Measurements will perform prior to ESWT,immidiately after the first ESWT and last ESWT treatment.Change of fiber length in 3 weeks
  'Logiq s7 Expert' US device including b-flow, semi-quantification and elastography, flow quantification, contrast imaging, b-steer and volume imaging device and with 11 L-D linear volume convex and linear probe will use for the measurements. During the evaluation, the muscles will place in the most relaxed position and no contraction will request. Fiber length will measure as the length of the fascicular path between the superficial and deep aponeurosis. For the measuring of the fiber length , the most clearly measure areas will be taken into consideration. If the fascicle extended off the image, the missing portion will estimate via linear extrapolation of the fascicle and aponeurosis
muscle thickness | Measurements will perform prior to ESWT,immidiately after the first ESWT and last ESWT treatment.Change of thickness in 3 weeks
  'Logiq s7 Expert' US device including b-flow, semi-quantification and elastography, flow quantification, contrast imaging, b-steer and volume imaging device and with 11 L-D linear volume convex and linear probe will use for the measurements. During the evaluation, the muscles will place in the most relaxed position and no contraction will reques thickness will measure in transversal as the distance between the superficial and the deep fascia at distance

SECONDARY OUTCOMES:
Quadriceps muscle flexibility | Measurements will perform prior to ESWT,immidiately after the first ESWT and last ESWT treatment.Change of flexibility in 3 weeks
  The Ely's test will use for the measurement. The procedure will modify to incorporate active knee ﬂexion (rather than passive knee ﬂexion) into the testing protocol in order to facilitate goniometer measurement by only one examiner. Participants will instruct to actively ﬂex one knee and bring their heel towards the buttocks, while maintaining a neutral pelvic posture and contact of the anterior aspect of the hip with the plinth.Goniometric scores will be taken in degrees
Hamstring muscle flexibility | Measurements will perform prior to ESWT,immidiately after the first ESWT and last ESWT treatment..Change of flexibility in 3 weeks
  Flexibility of the muscles will be measured with using tape measure. A single measurement will be performed for each muscle. The muscle flexibility will record as centimeters (cm).The passive straight leg raise (PSLR) test will perform to assess the hamstring muscle flexibility. The subjects will lay supine with their legs will straight on an examining bed. The ankle of the testing leg will keep in a relaxed position throughout testing. The endpoint for the PSLR test will determine by the following two criteria: (i) the tightness felt by the examiner and (ii) the onset of pain in the hamstring reported by subject. Evaluation will do according to the angle on the hip. The scores will measure by tape measure. The distance between calcaneus and the floor will record.
Gastrocinemius muscle flexibility | Measurements will perform prior to ESWT,immidiately after the first ESWT and last ESWT treatment..Change of flexibility in 3 weeks
  The lunge test will use for gastrocinemius. The patient will stand against the wall so that the distance between the foot and the wall is about 10 cm long. They will move one foot back a foot's distance behind the other.
  They will bend the front knee until it will touch the wall (keeping the heel on ground).
  If knee can not touch wall without heel coming off ground, the foot will be moved closer to wall and then will be repeated.
  If knee can touch wall without heel coming off ground, the foot will be moved further away from wall and then will be repeated.
  Keep will be repeated step 5 until can just touch knee to wall and heel stays on ground.The flexion lunge will be measured the distance length in centimeters (to the nearest O.lcm) from the end of the big toe to the wall using a tape measure on the floor .
Quadriceps muscle strength | Measurements will perform prior to ESWT,immidiately after the first ESWT and last ESWT treatment..Change of strength in 3 weeks
  Powertrak Hand-Held Dynamometer (JTech Medical, Utah, USA) digital dynamometer will use for assessing the muscle strength.The muscle strength will record as Newtons.Providing verbal encouragement to use their maximum efforts, the patients will ask to apply forces to the dynamometer during a period of 5 to 10 seconds while patients will sitting in a fixed chair and the examiner's hand pressed down the thigh to the chair.
hamstring muscle strength | Measurements will perform prior to ESWT,immidiately after the first ESWT and last ESWT treatment. Change of strength in 3 weeks
  Powertrak Hand-Held Dynamometer (JTech Medical, Utah, USA) digital dynamometer will use for assessing the muscle strength.The muscle strength will record as Newtons.. For the hamstring muscle, isometric knee flexion strength will measure with the subject in a prone position and the pelvis and the contralateral leg will be fixed. The dynamometer will place at the ankle, perpendicular to the lower leg. The foot will in plantar flexion and the knee in an extended position. Three maximal voluntary isometric knee flexion contractions will ask with gradually increasing effort
gastrokinemius muscle strength | Measurements will perform prior to ESWT,immidiately after the first ESWT and last ESWT treatment.Change of strength in 3 weeks
  Powertrak Hand-Held Dynamometer (JTech Medical, Utah, USA) digital dynamometer will use for assessing the muscle strength.The muscle strength will record as Newtons. All subjects will be performed the isometric contractions in a prone position on the table with the hip and knee extended and the foot in neutral position.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Private Hatem Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atamaz F, Ozcaldiran B, Ozdedeli S, Capaci K, Durmaz B. Interobserver and intraobserver reliability in lower-limb flexibility measurements. J Sports Med Phys Fitness. 2011 Dec;51(4):689-94. PMID 22212274
- [Background] Shechtman O, Gestewitz L, Kimble C. Reliability and validity of the DynEx dynamometer. J Hand Ther. 2005 Jul-Sep;18(3):339-47. doi: 10.1197/j.jht.2005.04.002. PMID 16059855
- [Background] English C, Fisher L, Thoirs K. Reliability of real-time ultrasound for measuring skeletal muscle size in human limbs in vivo: a systematic review. Clin Rehabil. 2012 Oct;26(10):934-44. doi: 10.1177/0269215511434994. Epub 2012 Feb 9. PMID 22324054
- [Background] Strasser EM, Draskovits T, Praschak M, Quittan M, Graf A. Association between ultrasound measurements of muscle thickness, pennation angle, echogenicity and skeletal muscle strength in the elderly. Age (Dordr). 2013 Dec;35(6):2377-88. doi: 10.1007/s11357-013-9517-z. Epub 2013 Mar 2. PMID 23456136
- [Background] Valle MS, Casabona A, Micale M, Cioni M. Relationships between Muscle Architecture of Rectus Femoris and Functional Parameters of Knee Motion in Adults with Down Syndrome. Biomed Res Int. 2016;2016:7546179. doi: 10.1155/2016/7546179. Epub 2016 Nov 8. PMID 27896273
- [Background] Vetrano M, d'Alessandro F, Torrisi MR, Ferretti A, Vulpiani MC, Visco V. Extracorporeal shock wave therapy promotes cell proliferation and collagen synthesis of primary cultured human tenocytes. Knee Surg Sports Traumatol Arthrosc. 2011 Dec;19(12):2159-68. doi: 10.1007/s00167-011-1534-9. Epub 2011 May 27. PMID 21617986
- [Background] Kim YW, Chang WH, Kim NY, Kwon JB, Lee SC. Effect of Extracorporeal Shock Wave Therapy on Hamstring Tightness in Healthy Subjects: A Pilot Study. Yonsei Med J. 2017 May;58(3):644-649. doi: 10.3349/ymj.2017.58.3.644. PMID 28332373
- [Background] Erroi D, Sigona M, Suarez T, Trischitta D, Pavan A, Vulpiani MC, Vetrano M. Conservative treatment for Insertional Achilles Tendinopathy: platelet-rich plasma and focused shock waves. A retrospective study. Muscles Ligaments Tendons J. 2017 May 10;7(1):98-106. doi: 10.11138/mltj/2017.7.1.098. eCollection 2017 Jan-Mar. PMID 28717617
- [Background] Zwerver J, Verhagen E, Hartgens F, van den Akker-Scheek I, Diercks RL. The TOPGAME-study: effectiveness of extracorporeal shockwave therapy in jumping athletes with patellar tendinopathy. Design of a randomised controlled trial. BMC Musculoskelet Disord. 2010 Feb 8;11:28. doi: 10.1186/1471-2474-11-28. PMID 20144188
- [Background] Askling C, Saartok T, Thorstensson A. Type of acute hamstring strain affects flexibility, strength, and time to return to pre-injury level. Br J Sports Med. 2006 Jan;40(1):40-4. doi: 10.1136/bjsm.2005.018879. PMID 16371489
- [Background] Ozbek EA, Kalem M, Kinik H. Do the Loss of Thigh Muscle Strength and Tibial Malrotation Cause Anterior Knee Pain after Tibia Intramedullary Nailing? Biomed Res Int. 2019 Mar 27;2019:3072105. doi: 10.1155/2019/3072105. eCollection 2019. PMID 31032341
- [Background] Arya S, Kulig K. Tendinopathy alters mechanical and material properties of the Achilles tendon. J Appl Physiol (1985). 2010 Mar;108(3):670-5. doi: 10.1152/japplphysiol.00259.2009. Epub 2009 Nov 5. PMID 19892931
- [Background] Miyamoto N, Hirata K, Kimura N, Miyamoto-Mikami E. Contributions of Hamstring Stiffness to Straight-Leg-Raise and Sit-and-Reach Test Scores. Int J Sports Med. 2018 Feb;39(2):110-114. doi: 10.1055/s-0043-117411. Epub 2017 Nov 30. PMID 29190853
- [Background] Massey G, Evangelidis P, Folland J. Influence of contractile force on the architecture and morphology of the quadriceps femoris. Exp Physiol. 2015 Nov;100(11):1342-51. doi: 10.1113/EP085360. Epub 2015 Oct 14. PMID 26374174
- [Background] Turton P, Hay R, Taylor J, McPhee J, Welters I. Human limb skeletal muscle wasting and architectural remodeling during five to ten days intubation and ventilation in critical care - an observational study using ultrasound. BMC Anesthesiol. 2016 Nov 29;16(1):119. doi: 10.1186/s12871-016-0269-z. PMID 27894277
- [Background] Karagiannidis E, Kellis E, Galanis N, Vasilios B. Semitendinosus muscle architecture during maximum isometric contractions in individuals with anterior cruciate ligament reconstruction and controls. Muscles Ligaments Tendons J. 2017 May 10;7(1):147-151. doi: 10.11138/mltj/2017.7.1.147. eCollection 2017 Jan-Mar. PMID 28717622
- [Background] Peeler J, Anderson JE. Reliability of the Ely's test for assessing rectus femoris muscle flexibility and joint range of motion. J Orthop Res. 2008 Jun;26(6):793-9. doi: 10.1002/jor.20556. PMID 18186129
- [Background] Bennell KL, Talbot RC, Wajswelner H, Techovanich W, Kelly DH, Hall AJ. Intra-rater and inter-rater reliability of a weight-bearing lunge measure of ankle dorsiflexion. Aust J Physiother. 1998;44(3):175-180. doi: 10.1016/s0004-9514(14)60377-9. PMID 11676731